CLINICAL TRIAL: NCT05572762
Title: A Prospective Comparative Study Between an Atraumatic Peribulbar Block and the Traditional Peribulbar Needle Technique
Brief Title: Assessing the Atraumatic Technique in Ophthalmic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Dina Moustafa Mohamed, Researcher of Anesthesia- Research Institute of Ophthalmology, Research Institute of Ophthalmology, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-3-27-5-2
Record Dates: First submitted 2022-07-10; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Intravenous Cannula Regional Ophthalmic Anesthesia

STUDY DESIGN:
Who Masked: Participant
Masking Description: the participant is going to have regional ophthalmic anesthesia, by either the atraumatic or the needle technique without being informed by which technique he is going to receive the block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic Peribulbar Technique (Experimental): a cannula is used to apply ophthalmic block
  Interventions: Device: Cannula plastic part while applying peribulbar block
- Conventional peribulbar block (Active Comparator): a 24 or 25 gauge needle is used to provide regional o anesthesia to the study group
  Interventions: Procedure: traditional technique

INTERVENTIONS:
Device: Cannula plastic part while applying peribulbar block — Using the cannula and introducing it peribulbar to apply regional ophthalmic anesthesia avoiding by this causing trauma to the globe, as the normal globe consistency is marble-like, the cannula can't puncture except in case of presence of staphyloma, so the cannula will either curve around it or will be kinked causing failure of the technique.
  Other Names: Atraumatic peribulbar technique
  Arms: Atraumatic Peribulbar Technique
Procedure: traditional technique — the patients are going to receive the local anesthetic standard of care technique by using 23- or 24-gauge needle introduced through the skin extra-conal and local anesthetic solution will be injected with volume AND concentration according to the surgery going to be done
  Other Names: needle traumatic peribulbar anesthesia
  Arms: Conventional peribulbar block

SUMMARY:
This study is conducted to determine the efficacy of the cannula atraumatic technique as an alternative to the traditional needle penetrating technique to minimize the incidence of accidental globe penetration and/ or perforation, as the plastic part of the cannula is blunt and is difficult to perforate the normal globe being marble-like in consistency.

DETAILED DESCRIPTION:
A prospective comparative single blinded randomized controlled clinical study was held in the operating theatre at Research institute of ophthalmology, on adult patients with age group between 18- 80 years of both sexes undergoing anterior, posterior segment or plastic surgeries. two techniques were used in comparison: the atraumatic technique, using a 20 or 22-gauge cannula advanced in the inferior-temporal peribulbar space after local infiltration. The skin and the conjunctiva will be pierced by the cannula and advanced for only 0.5 cm, then the cannula will be advanced blindly. Supplementation using the other sites (medial canthus and superior nasal) as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Both
3. patients going to do anterior, posterior segment surgery or cornea surgeries.

Exclusion Criteria:

1. Pediatric population
2. Mentally retarded patients
3. Patients having Problems to lie flat, refused to take regional
4. Patients with communication problems as; language barrier, deaf and mute.
5. Patients with bleeding diathesis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Safe Ophthalmic block using Globe Akinesia Score by Sarvela | 3 years
  A scoring system out of 12 to assess the four recti muscles, orbicularis oculi and the levator palpebri superioris degree of akinesia post regional anesthesia where 2 is full movement 0 is total block, and also the anesthesia is assessed where 2 is full sensation and 0 is considered total anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Ophthalmology, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
only the results